CLINICAL TRIAL: NCT02549599
Title: Chat/Text Program: Digital Health Information Efficacy Trial
Brief Title: Evaluating a Digital Health Information Tool
Acronym: Chat/Text
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: Planned Parenthood Federation of America (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Chat/Text Program
Record Dates: First submitted 2015-09-10; First posted 2015-09-15 (Estimated); Last update posted 2022-10-27 (Actual); Status verified 2017-09

CONDITIONS: Behavior and Behavior Mechanisms
Keywords: Digital and mobile health; Sexual and reproductive health; Adolescents and young adults
MeSH Terms: conditions — Behavior; Coitus | interventions — Treatment Delay

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Delayed Treatment (Other): Participants will receive a baseline survey and be routed to the Planned Parenthood website. No subsequent survey will be administered.
  Interventions: Other: Delayed Treatment
- Chat/Text Program (Experimental): Participants will receive real-time answers to questions they have about sexual and reproductive health topics from trained chat agents via the digital intervention program.
  Interventions: Behavioral: Chat/Text Program
- Website Content (Other): Participants will be routed to the Planned Parenthood website to information and content about issues regarding sexual and reproductive health.
  Interventions: Behavioral: Website Content

INTERVENTIONS:
Behavioral: Chat/Text Program — Participants will receive access to the Chat/Text program on the internet via computer or mobile device. The Chat/Text program involves interactive, immediate, and tailored messages (with pre-determined content) delivered by Chat/Text agents via online chat or mobile phone text. At the conclusion of the session, the participants will receive a combination-baseline and follow-up survey.
  Arms: Chat/Text Program
Behavioral: Website Content — Participants will be directed to content and information on the Planned Parenthood website. The website contains information on birth control methods, locations of Planned Parenthood health clinics, and on sexual and reproductive health more broadly.
  Arms: Website Content
Other: Delayed Treatment — Participants will receive a baseline survey and be routed to the Planned Parenthood website. No subsequent survey will be administered
  Arms: Delayed Treatment

SUMMARY:
The primary aim of the proposed project is to conduct a randomized controlled trial to evaluate the efficacy of a digital intervention tool that enables young people to correspond with trained staff via online chat or text messages about urgent questions related to sexual/reproductive health.

DETAILED DESCRIPTION:
The present evaluation study engages digital technology to target young people to impact their use of sexual health services. The primary aim of the proposed project is to conduct a randomized controlled trial to evaluate the efficacy of an intervention tool that enables young people to correspond with trained staff via online chat or text messages about urgent questions related to sexual/reproductive health. Specifically, Chat/Text is a program designed to provide immediate answers to urgent sexual and reproductive health questions from a reliable and confidential source and to link young people to sexual and reproductive health services. Agents are trained on substantive topics, and on responding compassionately and appropriately. They are provided scripted responses to specific topics. Agent performance is monitored and evaluated to ensure high-quality responses that meet the goals of the program. The program targets groups experiencing sexual and reproductive health disparities, particularly Black and Latino/Hispanic teens and young adults. The Chat/Text program was launched in September 2010 by Planned Parenthood Federation of America (PPFA). The present project is evaluating the efficacy of the Chat/Text program. Specifically, the investigators will compare the effect of the Chat/Text program to the standard of care available from PPFA (website content) in the absence of the Chat/Text program.

Participants will be randomized into one of the three arms of the evaluative study (experimental, control, and passive control). Participants in the experimental arm will receive access to the digital Chat/Text program where they can ask questions and receive answers about sexual and reproductive health issues in real-time, immediately followed by a combined baseline and follow-up assessment. Participants in the control arm of the study will be routed to the Planned Parenthood website to content and information on sexual and reproductive health issues, also followed by the combined assessment. Participants in the passive control will receive a standalone baseline assessment and then be routed to the website. No additional contact will be made with the passive control group.

The experimental participants will receive booster sessions in the form of e-mail and SMS communications. The first (5 days post-intervention) and second (3 weeks post-intervention) booster sessions will focus on appointment adherence. The third (2 months post-intervention) and fourth (2.5 months post-intervention) booster sessions will focus on effective birth control methods in addition to appointment adherence.

The control condition will not receive booster sessions, but will receive communications that aim to obtain additional tracking information. These tracking communications will be sent at the same time points as the experimental booster sessions (i.e., 5 days-, 3 weeks-, 2 months-, and 2.5 months-post website exposure).

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 15-25
* Had sex within the past 30 days prior to enrollment
* Never used the Planned Parenthood Chat/Text program

Exclusion Criteria:

* Males
* Females outside the ages of 15-25
* Female who report not having sex in the past 30 days
* Have used the Planned Parenthood Chat/Text program

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5220 (Actual)
Dates: Start 2015-02; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Increasing clinic attendance | Measured at 10 days post-intervention
  Increasing clinic attendance is measured using a self-report item that indicates if a participant completed a clinic appointment.
Increasing clinic attendance | Measured at 30 days post-intervention
  Increasing clinic attendance is measured using a self-report item that indicates if a participant completed a clinic appointment.
Increasing clinic attendance | Measured at 3 months post-intervention
  Increasing clinic attendance is measured using a self-report item that indicates if a participant completed a clinic appointment.

SECONDARY OUTCOMES:
Use of more effective birth control use | Measured at 10 days post-intervention
  The use of more effective birth control use is determined, through a self-report question asking if a participant changed her method of birth control to a more effective one. For example, a participant may change from a barrier method (e.g., condom) to a hormonal method.
Use of more effective birth control use | Measured at 30 days post-intervention
  The use of more effective birth control use is determined, through a self-report question asking if a participant changed her method of birth control to a more effective one. For example, a participant may change from a barrier method (e.g., condom) to a hormonal method.
Use of more effective birth control use | Measured at 3 months post-intervention
  The use of more effective birth control use is determined, through a self-report question asking if a participant changed her method of birth control to a more effective one. For example, a participant may change from a barrier method (e.g., condom) to a hormonal method.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Guilamo-Ramos, PhD, MPH, LCSW, RN, Principal Investigator — New York University; Leslie Kantor, PhD, MPH, Principal Investigator — Planned Parenthood Federation of America; James Jaccard, PhD, Principal Investigator — New York University
Locations (1):
- Planned Parenthood Federation of America, New York, New York, United States

REFERENCES:
- See also: Website Content Information — http://www.plannedparenthood.org/